CLINICAL TRIAL: NCT00706628
Title: A Multi-centre 3-arm Randomised Phase II Trial of BIBF 1120 Versus BIBW 2992 Versus Sequential Administration of BIBF 1120 and BIBW 2992 in Patients With Hormone-resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1239.3
Record Dates: First submitted 2008-06-24; First posted 2008-06-27 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — nintedanib; Afatinib

INTERVENTIONS:
Drug: BIBF 1120
Drug: BIBW 2992
Drug: Sequential BIBF 1120 + BIBW 2992

SUMMARY:
The primary objective of this trial is to estimate and compare the 12-week progression-free rate of BIBF 1120, BIBW 2992 or sequential administration of BIBF 1120 and BIBW 2992 in patients with HRPC as determined by radiographic, bone and PSA criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Signed informed consent.
* Able to comply with protocol requirements.
* Histologically, cytologically or biochemically documented adenocarcinoma of the prostate, clinically refractory or resistant to hormone therapy, as documented by progression following at least one hormonal therapy, which must include orchidectomy or gonadotropin releasing hormone agonist (GnRHa).
* Progressive Disease (PD) is defined as a minimum of three consecutive serum PSA measurements obtained at least 7 days apart within the previous 3 months of start of trial, which document progressively increasing values. Patients with progression of measurable disease (RECIST) or progression of bone disease must also fit the criterion for PSA progression.
* Patients must have documented progression (as defined above) following anti-androgen withdrawal of 4 weeks duration for flutamide and 6 weeks for bicalutamide or nilutamide. For a patient who has withdrawn from anti-androgen therapy less than 6 months prior to inclusion in trial one of the following criteria is also required:
* Following the completion of the anti-androgen withdrawal period one PSA higher than the last pre-withdrawal PSA.
* Or Following the completion of the anti-androgen withdrawal period if the PSA value has decreased, he can still qualify if 2 increases in PSA are documented after the post- withdrawal nadir.
* PSA > 5ng/mL.
* Life expectancy of at least 12 weeks.
* ECOG performance status 0-1 (see appendix 11.2).
* Stable analgesia requirements.
* Adequate hepatic function: total bilirubin < 26µmol/L, ALT and/or AST < 1.5x upper limit of normal (ULN).
* Adequate renal function: serum creatinine < 1.5 x ULN.
* INR Prothrombin time (PT) and partial thromboplastin time (PTT) <1.5 upper limit of normal.
* Absolute neutrophil count (ANC) > 1.5 x 109l, Platelets > 100 x 109/l.
* Haemoglobin > 9.0 g/dl.
* LVEF > 50 % on MUGA scan or echocardiogram.
* Castrate testosterone level [< 20ng/dl or <0.69nM (nM/L x 28.8 = ng/dl)], which must be maintained during the duration of the trial by orchidectomy or medical castration.
* Patient on oral or intravenous bisphosphonates are allowed to enter the trial as long as they have been on bisphosphonates for a minimum of 3 months.

Exclusion Criteria:

* Prior treatment with inhibitors of EGFR, HER 2 and/or VEGF receptors.
* Prior treatment with cytotoxic chemotherapy.
* Known hypersensitivity to the trial drugs or their excipients.
* Systemic corticosteroids 28 days before screening (inhaled corticosteroids prescribed for bronchospasm are allowed). Patients on long-term stable-dose steroids for concurrent illness are not excluded.
* Treatment with any investigational drug within 28 days of trial onset.
* History of other malignancies which could affect compliance with the protocol or interpretation of results within 5-years. Patients with adequately treated basal or squamous cell skin cancer are generally eligible.
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or active ulcers (gastro-intestinal tract, skin) or laboratory abnormality that may increase the risk associated with trial participation or trial drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the trial.
* Major injuries and/or surgery within 4 weeks of trial onset or bone fracture and planned surgical procedures during the trial period.
* Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within past 9 months, congestive heart failure > NYHA II) (see appendix 11.5).
* History of haemorrhagic or thrombotic event in the past 12 months. Known inherited predisposition to bleeds or to thrombosis.
* Patient with history or clinical evidence of CNS disease or brain metastases.
* Patients with symptoms of impending or established spinal cord compression.
* Gastrointestinal disorders or abnormalities that would inhibit absorption of the trial drug.
* Patients who require full-dose anticoagulation.
* Radio- or immunotherapy within the past four weeks prior to treatment with the trial drug.
* Patients unable to comply with the protocol.
* Active alcohol or drug abuse.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2006-03; Primary Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (9):
- United Kingdom (9):
  - 1239.3.4402 Boehringer Ingelheim Investigational Site, Belfast
  - 1239.3.4406 Boehringer Ingelheim Investigational Site, Bournemouth
  - 1239.3.4408 Boehringer Ingelheim Investigational Site, Brighton
  - 1239.3.4409 Boehringer Ingelheim Investigational Site, Cheltenham
  - 1239.3.4405 Boehringer Ingelheim Investigational Site, Glasgow
  - 1239.3.4403 Boehringer Ingelheim Investigational Site, Newcastle upon Tyne
  - 1239.3.4411 Boehringer Ingelheim Investigational Site, Southampton
  - 1239.3.4401 Boehringer Ingelheim Investigational Site, Sutton
  - 1239.3.4410 Boehringer Ingelheim Investigational Site, Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- BIBF 1120 Monotherapy: 250 mg soft gelatine capsules administered orally twice a day (BID). Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression.
- BIBW 2992 Monotherapy: 40 mg tablets administered orally once a day (QD). Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression.
- ComBI 40: Sequential alternating BIBF 1120 and BIBW 2992 combination therapy.
  Treatment regimen:
  BIBF 1120 250 mg BID on Days 1 to 7 and 15 to 21, BIBW 2992 40 mg QD on Days 8 to 14 and 22 to 28.
  Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression
- ComBI 70: Sequential alternating BIBF 1120 and BIBW 2992 combination therapy.
  Treatment regimen:
  BIBF 1120 250 mg BID on Days 1 to 7 and Days 15 to 21 of each treatment cycle; BIBW 2992 70 mg QD on Days 8 to 14 and Days 22 to 28 of each treatment cycle.
  The starting dose of BIBW 2992 was reduced due to an unexpectedly high incidence of severe (Grade 3) Adverse Events (AE) reported for the first 3 patients treated with ComBI 70. As the reported Adverse Events were attributed to BIBW 2992, the starting dose of BIBW 2992 in subsequent patients in this treatment arm was reduced to 40mg QD (ComBI 40); the dose of BIBF 1120 remained unchanged.
  Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression.
Period: Overall Study
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70
Started | 47 | 21 | 16 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 47 | 21 | 16 | 3
Not completed — Other Adverse Event | 16 | 5 | 5 | 2
Not completed — Non compliant with protocol | 0 | 1 | 0 | 0
Not completed — Consent withdrawn | 6 | 1 | 3 | 0
Not completed — Progressive disease | 20 | 13 | 8 | 1
Not completed — Other than those stated above | 4 | 0 | 0 | 0
Not completed — Not treated | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: The Treated Set consisted of all patients who received at least 1 dose of study medication.
Groups:
- ComBI 70: Sequential alternating BIBF 1120 and BIBW 2992 combination therapy.
  Treatment regimen:
  BIBF 1120 250 mg BID on Days 1 to 7 and Days 15 to 21 of each treatment cycle; BIBW 2992 70 mg QD on Days 8 to 14 and Days 22 to 28 of each treatment cycle.
  The starting dose of BIBW 2992 was reduced due to an unexpectedly high incidence of severe (Grade 3) Adverse Events reported for the first 3 patients treated with ComBI 70. As the reported Adverse Events were attributed to BIBW 2992, the starting dose of BIBW 2992 in subsequent patients in this treatment arm was reduced to 40mg QD (ComBI 40); the dose of BIBF 1120 remained unchanged.
  Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression.
- Total: Total of all reporting groups
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70 | Total
Number analyzed (Participants) | 46 | 20 | 16 | 3 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.7 (8.1) | 68.4 (5.4) | 70.4 (8.1) | 68.3 (0.6) | 68.4 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 46 | 20 | 16 | 3 | 85

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Rate (PFR) at 12 Weeks
Description: PFR is defined as a composite endpoint for disease progression.
  If patients met one of the following criteria they were counted as having progressive disease (PD):
  * Prostate serum antigen (PSA) progression according to Prostate-Specific Antigen Working Group (PSAWG) criteria
  * Bone metastasis progression- development of new lesions on bone scan or development of disease-related skeletal related events (SREs)
  * Disease progression according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.0
Time Frame: 12 weeks
Population: Modified full analysis set(mFAS): Patients who received at least 1 dose of study medication and for whom progression status could be determined at 12 weeks,excluding patients who discontinued treatment before 12 weeks for reasons other than PD.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70
Number analyzed (Participants) | 27 | 12 | 10 | 1
percentage of participants | 25.9 [13.17 to 44.68] | 0.0 [0.00 to 24.25] | 0.0 [0.00 to 27.75] | NA [NA to NA] — Not calculated to avoid reporting patient level data as only 1 patient had evaluable data
Statistical Analysis 1: Comparison: BIBF 1120 Monotherapy vs BIBW 2992 Monotherapy; Test type: Superiority or Other; p = 0.0577, Fisher Exact
Statistical Analysis 2: Comparison: BIBF 1120 Monotherapy vs ComBI 40; Test type: Superiority or Other; p = 0.0863, Fisher Exact

2. Secondary Outcome: Progression Free Rate at 24 and 48 Weeks
Description: PFR is defined as a composite endpoint for disease progression.
  If patients met one of the following criteria they were counted as having progressive disease (PD):
  * Prostate serum antigen (PSA) progression according to Prostate-Specific Antigen Working Group (PSAWG) criteria
  * Bone metastasis progression- development of new lesions on bone scan or development of disease-related skeletal related events (SREs)
  * Disease progression according to RECIST version 1.0
Time Frame: 24 weeks and 48 weeks
Population: Full analysis set (FAS), which consisted of all patients who received at least
  1 dose of study medication and for whom progression status could be determined at 12 weeks.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
percentage of participants
  24 weeks | 22.2 [10.61 to 40.76] | 0.0 [0.00 to 22.81] | 0.0 [0.00 to 27.75]
  48 weeks | 18.5 [8.18 to 36.70] | 0.0 [0.00 to 22.81] | 0.0 [0.00 to 27.75]

3. Secondary Outcome: Number of Patients Showing Prostate Serum Antigen (PSA) Response
Description: PSA response was evaluated according to the PSAWG guidelines. All patients achieving a fall in PSA of ≥50% from baseline (confirmed with a second value at least 4 weeks later) fulfilled the criteria for PSA response. The confirmatory value had to be at least 50% lower than the baseline value, but could be higher than the original drop in PSA (first PSA value).
  However, the confirmatory value could not be 50% higher than the first PSA value. If it was ≥50% higher than the first PSA, another sample was taken to determine if response had been achieved.
Time Frame: End of trial visit, 29 ± 1 days after Day 1 of the last treatment cycle (Up to 48 weeks)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
percentage of participants
  Response | 3.7 | 0.0 | 10.0
  No Response | 96.3 | 100.0 | 90.0
Statistical Analysis 1: Comparison: BIBF 1120 Monotherapy vs BIBW 2992 Monotherapy; Test type: Superiority or Other; Slope = 1.4823, 95% CI 2-sided [1.1754 to 1.7892], Standard Error of Mean 0.1490

4. Secondary Outcome: Duration of PSA Response
Description: Duration of PSA response was calculated from the time of first 50% decline in PSA (compared to baseline) until the time at which there was an increase of 50% from the PSA nadir, provided that the absolute increase was at least 5 ng/mL. The increase had to be confirmed by a second consecutive measurement that was at least 50% above the nadir. If the PSA never showed a 50% increase over the nadir value, then the patient was censored at the last PSA measurement.
  Duration of PSA response expressed in median number of days.
Time Frame: End of trial visit, 29 ± 1 days after Day 1 of the last treatment cycle (Up to 48 weeks)
Population: FAS
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- ComBI 40: Sequential alternating BIBF 1120 and BIBW 2992 combination therapy.
  Treatment regimen:
  BIBF 1120 250 mg BID on Days 1 to 7 and 15 to 21 BIBW 2992 40 mg QD on Days 8 to 14 and 22 to 28.
  Continuous daily dosing in 28-day cycles. Patients were eligible for repeated treatment cycles for 48 weeks in the absence of clinical disease progression
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
days | NA [NA to NA] — Not Applicable (NA) as only 1 patient had PSA response therefore the median and Inter-Quartile Range were not estimable using the Kaplan-Meier method. All other patients were censored. | NA [NA to NA] — NA as all patients censored | NA [NA to NA] — Not Applicable (NA) as only 1 patient had PSA response therefore the median and Inter-Quartile Range were not estimable using the Kaplan-Meier method. All other patients were censored.

5. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression through 48 weeks was calculated as the number of days from first administration of study drug to the first time that there was an increase of 50% from the PSA nadir, provided the absolute increase was at least 5 ng/mL.
  Time is expressed in median number of days.
Time Frame: Start of treatment until end of treatment (Up to 48 weeks)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
days | 31.0 [29.0 to 84.0] | 29.0 [29.0 to 57.0] | 57.0 [29.0 to 84.0]

6. Secondary Outcome: RECIST Tumour Progression Rate at 12, 24, 36, and 48 Weeks
Description: RECIST (version 1.0) tumour progression rate at 12, 24, 36, and 48 weeks was calculated based on the occurrence of new lesions, or an increase in the sum of the longest lesion diameters of at least 20%.
Time Frame: 12, 24, 36, and 48 weeks
Population: FAS (RECIST evaluable set); RECIST evaluable set, which consisted of patients who had RECIST measurable disease at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 12 | 8 | 7
percentage of participants
  12 weeks (N=12, 8, 7) | 8.3 | 50.0 | 42.9
  24 weeks (N=6, 1, 1) | 50.0 | 0.0 | 0.0
  36 weeks (N=3, 0, 0) | 33.3 | NA — Not Available (NA) as 0 participants analyzed | NA — NA as 0 participants analyzed
  48 weeks (N=2, 0, 0) | 50.0 | NA — NA as 0 participants analyzed | NA — NA as 0 participants analyzed

7. Secondary Outcome: Overall Objective Response by RECIST Criteria (Version 1.0) (Complete Response [CR] or Partial Response [PR]) for Patients With Measurable Disease at 12, 24, 36 and 48 Weeks
Description: Objective response is defined as a Complete or Partial response Complete response [CR] for Target lesions: Disappearance of all target lesions. Complete response [CR] for Non- target lesions: Disappearance of all non-target lesions and normalization of tumour marker level Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Time Frame: 12, 24, 36 and 48 weeks
Population: FAS (RECIST evaluable set)
Measure: Number; unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 12 | 8 | 7
percentage of participants
  12 weeks (N=12, 8, 7) | 8.3 | 0.0 | 0.0
  24 weeks (N=6, 1, 1) | 0.0 | 0.0 | 0.0
  36 weeks (N=3, 0, 0) | 0.0 | NA — Not Available (NA) as 0 participants analyzed | NA — NA as 0 participants analyzed
  48 weeks (N=2, 0, 0) | 0.0 | NA — NA as 0 participants analyzed | NA — NA as 0 participants analyzed

8. Secondary Outcome: Duration of RECIST Response
Description: Time from first observation of response (PR, CR, confirmed or unconfirmed) until progression according to RECIST (version 1.0) or death.
  Duration is expressed in Median number of days.
Time Frame: Up to 48 weeks
Population: FAS (RECIST evaluable set)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 12 | 8 | 7
days | 116.0 [116.0 to 116.0] | NA [NA to NA] — Not Applicable (NA) as 0 patients had RECIST response therefore the median and Inter-Quartile Range were not estimable using the Kaplan-Meier method. All patients were censored. | NA [NA to NA] — Not Applicable (NA) as 0 patients had RECIST response therefore the median and Inter-Quartile Range were not estimable using the Kaplan-Meier method. All patients were censored.

9. Secondary Outcome: Time to Progression
Description: Time from first administration of study drug until disease progression according to composite endpoint.
  Time is expressed in Median number of days.
Time Frame: start of treatment until end of the treatment (Up to 48 weeks)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
days | 31.0 [29.0 to 84.0] | 29.0 [29.0 to 54.0] | 57.0 [29.0 to 78.0]

10. Secondary Outcome: Overall Survival (Time to Death)
Description: Overall survival (time to death) was calculated in days from baseline to the date of reporting of death. Time is expressed in Median number of days.
Time Frame: start of treatment until 28 days after end of treatment (Up to 52 weeks)
Population: FAS
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40
Number analyzed (Participants) | 27 | 13 | 10
days | NA [NA to NA] — Not Applicable (NA) as all patients censored | NA [NA to NA] — NA as all patients censored | NA [NA to NA] — NA as all patients censored

11. Secondary Outcome: Incidence and Worst Intensity of Adverse Events With Grading According CTCAE
Description: Incidence and worst intensity of Adverse Events with grading according to the Common Terminology Criteria for Adverse Events (CTCAE version 3.0).
Time Frame: from first intake of treatment until 29 days after last intake of treatment (Up to 52 weeks)
Population: Treated Set
Measure: Number; unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70
Number analyzed (Participants) | 46 | 20 | 16 | 3
percentage of participants
  CTCAE Grade 1 | 26.1 | 0.0 | 37.5 | 0.0
  CTCAE Grade 2 | 30.4 | 55.0 | 18.8 | 33.3
  CTCAE Grade 3 | 37.0 | 40.0 | 37.5 | 66.7
  CTCAE Grade 4 | 6.5 | 0.0 | 0.0 | 0.0
  CTCAE Grade 5 | 0.0 | 5.0 | 6.3 | 0.0

12. Secondary Outcome: Changes in Safety Laboratory Parameters
Description: Changes in safety laboratory Parameters reported as adverse events
Time Frame: from first intake of treatment until 29 days after last intake of treatment (Up to 52 weeks)
Population: Treated Set
Measure: Number; unit: percentage of participants
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70
Number analyzed (Participants) | 46 | 20 | 16 | 3
percentage of participants
  Alanine aminotransferase increased | 17.4 | 5.0 | 18.8 | 33.3
  Gamma-glutamyltransferase increased | 4.3 | 0.0 | 12.5 | 33.3
  Aspartate aminotransferase increased | 10.9 | 0.0 | 18.8 | 0.0
  Blood urea increased | 2.2 | 10.0 | 0.0 | 0.0
  Blood creatinine increased | 2.2 | 5.0 | 0.0 | 0.0
  Blood potassium decreased | 0.0 | 5.0 | 0.0 | 0.0
  Transaminases increased | 4.3 | 0.0 | 0.0 | 0.0
  Blood alkaline phosphatase increased | 2.2 | 0.0 | 0.0 | 0.0
  Hepatic enzyme increased | 2.2 | 0.0 | 0.0 | 0.0

13. Secondary Outcome: Trough Plasma Concentrations for BIBF 1120 and BIBW 2992 for the Monotherapy
Description: Trough plasma concentrations are defined either as pre-dose concentration of BIBF 1120 and BIBW 2992 in plasma at steady state immediately before administration of the next dose for the monotherapy treatment or as post dose concentrations taken after the dosing interval for the combination treatment
Time Frame: Day 15, Day 29 and Day 57
Population: Pharmacokinetics (PK) data set: All patients from whom PK samples were received in the bioanalytical laboratories were included in the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy
Number analyzed (Participants) | 43 | 18
ng/mL
  Cpre,ss,15 (N=28, 15) | 10.2 (81.0) | 18.0 (81.2)
  Cpre,ss,29 (N=35, 18) | 11.8 (75.5) | 19.1 (92.6)
  Cpre,ss,57 (N=27, 12) | 11.8 (110.0) | 18.2 (81.5)

14. Secondary Outcome: Trough Plasma Concentrations for BIBF 1120 and BIBW 2992 for the Combination Therapy
Description: Trough plasma concentrations are defined either as pre-dose concentration of BIBF 1120 and BIBW 2992 in plasma at steady state immediately before administration of the next dose for the monotherapy treatment or as post dose concentrations taken after the dosing interval for the combination treatment (C12,14 for BIBF1120 ; C24,7 and C24,14 for BIBW2992)
  C12,14: plasma concentration at 12 hours Day 14
Time Frame: Day7, Day 14
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Combination Therapy of BIBF 1120 and BIBW 2992: Sequential alternating BIBF 1120 and BIBW 2992 combination therapy.
  C12,14 values of BIBF 1120 BS after sequential alternating 7-days administration of 250 mg BIBF 1120 bid;
  C24,7, C24,14 and C24,42 values of BIBW 2992 BS after sequential alternating 7-days administration of 40 mg BIBW 2992 qd
Arm/Group | Combination Therapy of BIBF 1120 and BIBW 2992
Number analyzed (Participants) | 16
ng/mL
  C 12,14 (N=14) | 13.7 (50.5)
  C 24,7 (N=13) | 11.4 (216)
  C 24,14 (N=12) | 16.4 (53.7)

ADVERSE EVENTS:
Time Frame: from first intake of treatment until 29 days after last intake of treatment (Up to 52 weeks)
Arm/Group | BIBF 1120 Monotherapy | BIBW 2992 Monotherapy | ComBI 40 | ComBI 70
Serious Adverse Events (participants affected / at risk) | 11/46 | 2/20 | 4/16 | 1/3
Other Adverse Events (participants affected / at risk) | 46/46 | 20/20 | 16/16 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 Monotherapy (N=46) | BIBW 2992 Monotherapy (N=20) | ComBI 40 (N=16) | ComBI 70 (N=3)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 2 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 Monotherapy (N=46) | BIBW 2992 Monotherapy (N=20) | ComBI 40 (N=16) | ComBI 70 (N=3)
Asthenopia (Eye disorders) | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 3 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 9 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 2 | 5 | 0
Diarrhoea (Gastrointestinal disorders) | 35 | 20 | 15 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 5 | 1 | 1
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 4 | 5 | 2
Nausea (Gastrointestinal disorders) | 29 | 5 | 6 | 2
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 5 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 16 | 4 | 4 | 2
Chest pain (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 7 | 9 | 3 | 3
Feeling drunk (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 2 | 0 | 0
Mucosal haemorrhage (General disorders) | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 0 | 0
Pain (General disorders) | 3 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 8 | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 3 | 0
Blood urea increased (Investigations) | 1 | 2 | 0 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram ST-T segment abnormal (Investigations) | 0 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 1 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 6 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 3 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 0 | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 4 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 3 | 4 | 1 | 1
Headache (Nervous system disorders) | 5 | 3 | 0 | 0
Lethargy (Nervous system disorders) | 9 | 5 | 7 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0
Affect lability (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 3 | 2 | 2 | 0
Nocturia (Renal and urinary disorders) | 6 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 2 | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 10 | 5 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 6 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 10 | 5 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 0 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Data from the ComBI 70 group were not included in analyses of efficacy, data was available for one patient for this group for the primary outcome however is not reported to avoid reporting patient level data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.